CLINICAL TRIAL: NCT05667077
Title: The Effect of Amantadine on Post-COVD-19 Fatigue: a Clinical Trial
Brief Title: The Effect of Amantadine on Post-COVD-19 Fatigue
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Ali Amini Harandi, Assistant Professor, Shahid Beheshti University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IR.SBMU.MSP.REC.1400.555
Record Dates: First submitted 2022-11-25; First posted 2022-12-28 (Actual); Last update posted 2022-12-28 (Actual); Status verified 2022-12

CONDITIONS: Post-COVID-19 Syndrome
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome | interventions — Amantadine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- amantadine (Experimental): The group that was treated with amantadine
  Interventions: Drug: Amantadine
- control (No Intervention): The group that was not treated

INTERVENTIONS:
Drug: Amantadine — The amantadine group is treated with amantadine capsules 100mg twice a day for two weeks
  Arms: amantadine

SUMMARY:
This study aimed to investigate amantadine's safety and its effect on reducing post-COVID-19 fatigue.

DETAILED DESCRIPTION:
Background The 2019 coronavirus disease has severely affected the health of the general public. Even after recovery, this disease can cause problems, including chronic fatigue, which the patient can suffer from for years and cause permanent disability for a number of patients.

Despite the fact that fatigue due to COVID-19 has affected many patients, not many studies have been done in the field of effective treatment for this problem.

In this study, the investigators studied the effect of amantadine on the fatigue of COVID-19 patients.

Method In this clinical trial study, 83 patients were randomly included in the study from the patients referred to the internal clinic of Shohada Tajrish Hospital in Tehran, and they were initially evaluated by VAFS and FSS questionnaires. 17 patients were initially excluded due to having at least one exclusion criterion. And 66 patients were randomly divided between two groups using amantadine and the control group. The amantadine group was treated with amantadine capsules 100 mg BD for 2 weeks and after 2 weeks again for both The group questionnaire was completed, and the data was analyzed by SPSS software version 26.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of COVID-19
* clinical evidence of fatigue despite the passage of 30 to 60 days from the onset --of the symptoms of COVID-19
* willingness and informed consent to participate in the study

Exclusion Criteria:

* the recurrence of COVID-19 in the form of re-infection
* history of psychiatric diseases
* psychotic disorders (in the form of hallucinations and delusions)
* anxiety disorders and major depression
* substance abuse in the last four months
* taking antidepressants during the last six weeks
* corticosteroids consumption during the last six weeks
* taking psychostimulant drugs
* an unstable medical condition
* cognitive disorders and confusion
* withdrawal from participating in the study
* history of rheumatological disease
* getting cancer and malignancy
* advanced chronic diseases (heart, liver, kidney, etc.)
* edema of organs
* hypertension (untreated)
* hypogonadism (untreated)
* hypothyroidism (untreated)
* anemia (untreated)
* pregnancy and breastfeeding
* nausea and vomiting when starting to take Amantadine
* convulsions
* dyspnea
* post-COVID-19 encephalopathy

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 83 (Estimated)
Dates: Start 2022-12-26 (Estimated); Primary Completion 2022-12-29 (Estimated); Study Completion 2023-01-10 (Estimated)

PRIMARY OUTCOMES:
Fatigue Severity Scale (FSS) | 2 weaks
  Comparison of fatigue scale score change before and after treatment with amantadine using FSS Minimum 1 Maximum 7 Higher score means greater fatique severity
Visual Analog Fatigue Scale (VAFS) | 2 weaks
  Comparison of fatigue scale score change before and after treatment with amantadine using VAFS Minimum 0 Maximum 100 Higher score means greater fatique severity

CONTACTS AND LOCATIONS:
Locations (1):
- Shohada Tajrish Hospital, Tehran, Iran

IPD SHARING:
Plan to Share IPD: No